CLINICAL TRIAL: NCT01690273
Title: Effect of Two Exercise Therapy Program With and Without Elastic Resistance in Ankylosing Spondylitis Patients
Brief Title: Exercise Therapy Program in Ankylosing Spondylitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Andrea Lopes Gallinaro, MASTER, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 8206212
Record Dates: First submitted 2012-09-18; First posted 2012-09-21 (Estimated); Results first posted 2016-10-20 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-08

CONDITIONS: Ankylosing Spondylitis
Keywords: exercise; mobility; strengthening; physiotherapy
MeSH Terms: conditions — Spondylitis, Ankylosing; Motor Activity | interventions — Range of Motion, Articular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ankylosing spondylitis control (No Intervention): control group
- mobility exercise (Experimental): mobility exercises
  Interventions: Other: mobility exercise
- mobility and elastic resistance exercise (Experimental): AS patients was submitted to a program mobility exercise plus elastic resistance exercises
  Interventions: Other: mobility and elastic resistance exercise

INTERVENTIONS:
Other: mobility exercise — 30 minutes, twice a week
  Arms: mobility exercise
Other: mobility and elastic resistance exercise — 30 minutes, twice a week each exercises group. (total 1 hour)
  Arms: mobility and elastic resistance exercise

SUMMARY:
Mobility exercises are used in Ankylosing Spondylitis (AS) patients to preserve and restore axial mobility, but there are no data regarding a specific rehabilitation program that includes flexibility alone and its association with resistance exercises in AS patients with stable disease activity. So, we assessed the effects of two exercise programs in terms of mobility, functional capacity, quality of life and disease activity in AS patients. Methods. Fifty-five sedentary AS patients with a Bath Ankylosing Spondylitis Activity Index (BASDAI) <4 were included.

DETAILED DESCRIPTION:
The AS patients were randomly assigned into three groups, to receive a mobility exercise program (M) or mobility plus elastic resistance exercise program (M+R) or no exercise (C). The exercises group sessions were conducted twice per week for 16 weeks. This supervised program comprised 30 minutes of outdoor stretching and mobility exercises for the spine and limbs (M). After the flexibility program, M+R group carry out more 30 minutes of elastic resistance exercises. The mobility, disease activity and functional parameters were evaluated at baseline and after 16 weeks, with the evaluator blinded to the treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Ankylosing spondylitis patient
* Basdai index lower than 4
* Physical inactive
* Functional class I to III

Exclusion Criteria:

* Fibromyalgia
* Cardiovascular disease
* Pain Visual Analogue Scale ("VAS") over 8

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Lucia Pinto, Phd, Study Chair — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
paper is been written

REFERENCES:
- [Result] Yigit S, Sahin Z, Demir SE, Aytac DH. Home-based exercise therapy in ankylosing spondylitis: short-term prospective study in patients receiving tumor necrosis factor alpha inhibitors. Rheumatol Int. 2013 Jan;33(1):71-7. doi: 10.1007/s00296-011-2344-6. Epub 2012 Jan 5. PMID 22218641

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two hundred nine consecutive patients from the division of rheumatology outpatient clinic of the university hospital (Clinics Hospital of University Medicine School of Sao Paulo) diagnosed with AS according to the modified New York criteria, were invited to participate. Fifty Five individuals were randomly allocated into three groups
Pre-assignment Details: Seventy patients did not accepted and 84 did not followed inclusion criteria. Fifty five were allocated into three groups after following the inclusion criteria.
Groups:
- Ankylosing Spondylitis Control: control group, no intervention in ankylosing spondylitis patients
- Mobility in Ankylosing Spondylitis: mobility exercises
  mobility exercise: 30 minutes, twice a week
- Mobility and Elastic Resistance Exercise in AS: mobility, plus elastic resistance exercises
  mobility and elastic resistance exercise: 30 minutes, twice a week each exercises group. (total 1 hour)
Period: Overall Study
Arm/Group | Ankylosing Spondylitis Control | Mobility in Ankylosing Spondylitis | Mobility and Elastic Resistance Exercise in AS
Started | 18 | 17 | 20
Completed | 18 | 17 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ankylosing Spondylitis Control: Following a randomization, patients from control group stays during sixteen weeks only with medical treatment.
- Stretching in AS: stretching exercises
  stretching exercise: 30 minutes, twice a week for sixteen weeks.
- Elastic Resistance Exercise in AS: stretching and elastic resistance exercises
  stretching and elastic resistance exercise: 30 minutes, twice a week each exercises group. (total 1 hour) for sixteen weeks.
- Total: Total of all reporting groups
Arm/Group | Ankylosing Spondylitis Control | Stretching in AS | Elastic Resistance Exercise in AS | Total
Number analyzed (Participants) | 18 | 17 | 20 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (10.8) | 49.2 (13.1) | 48.3 (11.1) | 48.2 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 7
  Male | 15 | 15 | 18 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 13 | 12 | 13 | 38
  More than one race | 5 | 5 | 7 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: FUNCTIONAL INDEX
Description: BASFI - Bath ankylosing spondylitis functional index. A scale from 0 to 10 (lower scores means better functional capacity), results are measured by mean and standard deviation.
Time Frame: Baseline and 16 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ankylosing Spondylitis Control: control group with AS patients and no exercise
- Mobility in AS: mobility exercises
  mobility exercise: 30 minutes, twice a week
- Mobility Plus Elastic Resistance Exercise in AS: mobility and elastic resistance exercises
  mobility and elastic resistance exercise: 30 minutes, twice a week each exercises group. (total 1 hour)
Arm/Group | Ankylosing Spondylitis Control | Mobility in AS | Mobility Plus Elastic Resistance Exercise in AS
Number analyzed (Participants) | 18 | 17 | 20
units on a scale
  baseline | 3.4 (2.7) | 4.3 (1.9) | 3.2 (2.6)
  16 weeks | 4.5 (2.5) | 4.0 (2.2) | 2.2 (2.0)
Statistical Analysis 1: Comparison: Ankylosing Spondylitis Control; Test type: Superiority or Other; p = 0.13, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mobility in AS; Test type: Superiority or Other; p = 0.99, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.11, Mixed Models Analysis
Statistical Analysis 4: Comparison: Ankylosing Spondylitis Control vs Mobility in AS; Test type: Superiority or Other; p = 0.9913, Mixed Models Analysis
Statistical Analysis 5: Comparison: Ankylosing Spondylitis Control vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.0427, Mixed Models Analysis
Statistical Analysis 6: Comparison: Mobility in AS vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.1856, Mixed Models Analysis

2. Primary Outcome: Mobility Index
Description: Bath ankylosing spondylitis motion index. A mean of five mobility measures committed by Ankylosing Spondylitis disease. Higher results means higher limitations in mobility (units of measure from 0 to 10)
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale from 0 to 10
Arm/Group | Ankylosing Spondylitis Control | Mobility in AS | Mobility Plus Elastic Resistance Exercise in AS
Number analyzed (Participants) | 18 | 17 | 20
units on a scale from 0 to 10
  baseline | 4.3 (2) | 5.3 (2) | 4.5 (2.1)
  16 weeks | 4.6 (2.0) | 4.8 (2.1) | 4.0 (2.1)
Statistical Analysis 1: Comparison: Ankylosing Spondylitis Control; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mobility in AS; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis
Statistical Analysis 4: Comparison: Ankylosing Spondylitis Control vs Mobility in AS; Test type: Superiority or Other; p = 1, Mixed Models Analysis
Statistical Analysis 5: Comparison: Ankylosing Spondylitis Control vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.935, Mixed Models Analysis
Statistical Analysis 6: Comparison: Mobility in AS vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.876, Mixed Models Analysis

3. Primary Outcome: Disease Activity Index
Description: BASDAI - Bath ankylosing spondylitis disease activity index. Scale from 0 to 6. Higher scores means worst disease activity. Numbers are expressed in average (SD)
Time Frame: Baseline and 16 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mobility in AS: mobility exercises
  mobility exercise: 30 minutes, twice a week for sixteen weeks.
- Mobility Plus Elastic Resistance Exercise in AS: mobility and elastic resistance exercises
  mobility and elastic resistance exercise: 30 minutes, twice a week each exercises group. (total 1 hour) for sixteen weeks.
Arm/Group | Ankylosing Spondylitis Control | Mobility in AS | Mobility Plus Elastic Resistance Exercise in AS
Number analyzed (Participants) | 18 | 17 | 20
units on a scale
  baseline | 2 (1) | 2.6 (1.1) | 2.1 (1.4)
  16 weeks | 3.2 (2.0) | 2.9 (1.4) | 1.7 (1.4)
Statistical Analysis 1: Comparison: Ankylosing Spondylitis Control; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mobility in AS; Test type: Superiority or Other; p = 0.87, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.83, Mixed Models Analysis
Statistical Analysis 4: Comparison: Ankylosing Spondylitis Control vs Mobility in AS; Test type: Superiority or Other; p = 0.989, Mixed Models Analysis
Statistical Analysis 5: Comparison: Ankylosing Spondylitis Control vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.022, Mixed Models Analysis
Statistical Analysis 6: Comparison: Mobility in AS vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.119, Mixed Models Analysis

4. Primary Outcome: Ankylosing Spondylitis Disease Activity Scale -Disease Activity
Description: Scores vary from 0 to 10, and higher than 4 scores are indicative of disease activity. Data are expressed by means and SD
Time Frame: Baseline and 16 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ankylosing Spondylitis Control: control group AS patients with no exercise
Arm/Group | Ankylosing Spondylitis Control | Mobility in AS | Mobility Plus Elastic Resistance Exercise in AS
Number analyzed (Participants) | 18 | 17 | 20
units on a scale
  baseline | 1.8 (0.7) | 1.7 (0.7) | 1.5 (0.7)
  16 weeks | 2.2 (0.8) | 1.6 (0.7) | 1.4 (0.7)
Statistical Analysis 1: Comparison: Ankylosing Spondylitis Control; Test type: Superiority or Other; p = 0.09, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mobility in AS; Test type: Superiority or Other; p = 0.99, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.94, Mixed Models Analysis
Statistical Analysis 4: Comparison: Ankylosing Spondylitis Control vs Mobility in AS; Test type: Superiority or Other; p = 0.213, Mixed Models Analysis
Statistical Analysis 5: Comparison: Ankylosing Spondylitis Control vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis
Statistical Analysis 6: Comparison: Mobility in AS vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.900, Mixed Models Analysis

5. Primary Outcome: Global Evaluation Self Reported
Description: Bath Ankylosing Spondylitis Global is a self reported global score varying from 0 to 10. Higher scores means worst health evaluation. Expressed by means and standard deviation.
Time Frame: Baseline and 16 Weeks
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Ankylosing Spondylitis Control | Mobility in AS | Mobility Plus Elastic Resistance Exercise in AS
Number analyzed (Participants) | 18 | 17 | 20
units on a scale
  baseline | 3.6 (1.9) | 5.0 (2.3) | 4.1 (2.6)
  16 weeks | 5.6 (2.4) | 4.7 (2.2) | 3.4 (2.5)
Statistical Analysis 1: Comparison: Ankylosing Spondylitis Control; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mobility in AS; Test type: Superiority or Other; p = 0.99, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.69, Mixed Models Analysis
Statistical Analysis 4: Comparison: Ankylosing Spondylitis Control vs Mobility in AS; Test type: Superiority or Other; p = 0.874, Mixed Models Analysis
Statistical Analysis 5: Comparison: Ankylosing Spondylitis Control vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.057, Mixed Models Analysis
Statistical Analysis 6: Comparison: Mobility in AS vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.526, Mixed Models Analysis

6. Secondary Outcome: Thoracolumbar Mobility
Description: Thoracolumbar rotation Pavelka. Measured with a tape in centimeters. Higher number means better thoracolumbar rotation
Time Frame: Baseline and 16 Weeks
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Ankylosing Spondylitis Control | Mobility in AS | Mobility Plus Elastic Resistance Exercise in AS
Number analyzed (Participants) | 18 | 17 | 20
Centimeters
  baseline | 1.9 (1.5) | 1.4 (0.9) | 1.6 (1.1)
  16 weeks | 1.7 (0.9) | 2.1 (1.0) | 2.6 (1.1)
Statistical Analysis 1: Comparison: Ankylosing Spondylitis Control; Test type: Superiority or Other; p = 0.853, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mobility in AS; Test type: Superiority or Other; p = 0.016, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.000, Mixed Models Analysis
Statistical Analysis 4: Comparison: Ankylosing Spondylitis Control vs Mobility in AS; Test type: Superiority or Other; p = 0.889, Mixed Models Analysis
Statistical Analysis 5: Comparison: Ankylosing Spondylitis Control vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.098, Mixed Models Analysis
Statistical Analysis 6: Comparison: Mobility in AS vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.645, Mixed Models Analysis

7. Secondary Outcome: Pain Scale
Description: Pain was evaluated in a visual analogue scale (VAS) from 0 to 10. higher scores means much pain. Data was expressed by means and standard deviation.
Time Frame: Baseline and 16 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ankylosing Spondylitis Control | Mobility in AS | Mobility Plus Elastic Resistance Exercise in AS
Number analyzed (Participants) | 18 | 17 | 20
units on a scale
  baseline | 1.8 (1.8) | 2.5 (1.9) | 2.0 (1.9)
  16 weeks | 2.3 (2.7) | 2.4 (1.5) | 2.0 (1.9)
Statistical Analysis 1: Comparison: Ankylosing Spondylitis Control; Test type: Superiority or Other; p = 0.07, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mobility in AS; Test type: Superiority or Other; p = 0.13, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.97, Mixed Models Analysis
Statistical Analysis 4: Comparison: Ankylosing Spondylitis Control vs Mobility in AS; Test type: Superiority or Other; p = 1, Mixed Models Analysis
Statistical Analysis 5: Comparison: Ankylosing Spondylitis Control vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.338, Mixed Models Analysis
Statistical Analysis 6: Comparison: Mobility in AS vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.476, Mixed Models Analysis

8. Secondary Outcome: Stiffness Scale
Description: Stiffness was measured by an VAS varying from 0 to 10. Higher scores means worst stiffness. Data are expressed by mean and SD.
Time Frame: Baseline and 16 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ankylosing Spondylitis Control | Mobility in AS | Mobility Plus Elastic Resistance Exercise in AS
Number analyzed (Participants) | 18 | 17 | 20
units on a scale
  baseline | 3.1 (2.6) | 3.1 (2.2) | 3.1 (2.4)
  16 weeks | 4.3 (2.6) | 4.2 (2.0) | 2.8 (2.0)
Statistical Analysis 1: Comparison: Ankylosing Spondylitis Control; Test type: Superiority or Other; p = 0.88, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mobility in AS; Test type: Superiority or Other; p = 0.99, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 1, Mixed Models Analysis
Statistical Analysis 4: Comparison: Ankylosing Spondylitis Control vs Mobility in AS; Test type: Superiority or Other; p = 1, Mixed Models Analysis
Statistical Analysis 5: Comparison: Ankylosing Spondylitis Control vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.995, Mixed Models Analysis
Statistical Analysis 6: Comparison: Mobility in AS vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.985, Mixed Models Analysis

9. Secondary Outcome: Short Form-12 (PCS)
Description: Quality of life was analyzed in a physical component score varying from 0 (lowest level of health) to 100 (highest level of health) scale. Data are expressed by mean and SD.
Time Frame: Baseline and 16 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ankylosing Spondylitis Control | Mobility in AS | Mobility Plus Elastic Resistance Exercise in AS
Number analyzed (Participants) | 18 | 17 | 20
units on a scale
  baseline | 42.3 (7.4) | 38.8 (8.0) | 43.9 (8.5)
  16 weeks | 41.9 (8.8) | 40.9 (10.6) | 44.8 (8.8)
Statistical Analysis 1: Comparison: Ankylosing Spondylitis Control; Test type: Superiority or Other; p = 0.9, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mobility in AS; Test type: Superiority or Other; p = 0.7, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.99, Mixed Models Analysis
Statistical Analysis 4: Comparison: Ankylosing Spondylitis Control vs Mobility in AS; Test type: Superiority or Other; p = 0.999, Mixed Models Analysis
Statistical Analysis 5: Comparison: Ankylosing Spondylitis Control vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.900, Mixed Models Analysis
Statistical Analysis 6: Comparison: Mobility in AS vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.739, Mixed Models Analysis

10. Secondary Outcome: Short Form-12 (MCS)
Description: Quality of life was analyzed in a mental component score varying from 0 (lowest level of health) to 100 (highest level of health). Data are expressed by mean and SD.
Time Frame: Baseline and 16 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ankylosing Spondylitis Control | Mobility in AS | Mobility Plus Elastic Resistance Exercise in AS
Number analyzed (Participants) | 18 | 17 | 20
units on a scale
  baseline | 51.8 (10.7) | 45.7 (11.6) | 47.1 (13.5)
  16 weeks | 52.1 (9.7) | 46.0 (10.8) | 51.6 (12.4)
Statistical Analysis 1: Comparison: Ankylosing Spondylitis Control; Test type: Superiority or Other; p = 1, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mobility in AS; Test type: Superiority or Other; p = 1, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.37, Mixed Models Analysis
Statistical Analysis 4: Comparison: Ankylosing Spondylitis Control vs Mobility in AS; Test type: Superiority or Other; p = 0.618, Mixed Models Analysis
Statistical Analysis 5: Comparison: Ankylosing Spondylitis Control vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 1, Mixed Models Analysis
Statistical Analysis 6: Comparison: Mobility in AS vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.689, Mixed Models Analysis

11. Secondary Outcome: MASES
Description: Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) score varying from 0 to 13. Where 0 is no painful point reported and 13 is all tender points reported as painful. Data are expressed by means and standard deviation
Time Frame: Baseline and 16 Weeks
Measure: Mean (Standard Deviation); unit: Number of painful tender points
Arm/Group | Ankylosing Spondylitis Control | Mobility in AS | Mobility Plus Elastic Resistance Exercise in AS
Number analyzed (Participants) | 18 | 17 | 20
Number of painful tender points
  baseline | 0.7 (1.4) | 1.5 (3.4) | 0.8 (1.7)
  16 weeks | 1.3 (1.9) | 1.1 (1.7) | 0.7 (1.5)
Statistical Analysis 1: Comparison: Ankylosing Spondylitis Control; Test type: Superiority or Other; p = 0.8, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mobility in AS; Test type: Superiority or Other; p = 0.97, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.99, Mixed Models Analysis
Statistical Analysis 4: Comparison: Ankylosing Spondylitis Control vs Mobility in AS; Test type: Superiority or Other; p = 0.999, Mixed Models Analysis
Statistical Analysis 5: Comparison: Ankylosing Spondylitis Control vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.929, Mixed Models Analysis
Statistical Analysis 6: Comparison: Mobility in AS vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.980, Mixed Models Analysis

12. Secondary Outcome: Chin-coronoid Distance
Description: lateral rotation of the head (chin-coronoid distance) was measured with a tape in centimeters. Highest score means better lateral rotation mobility. Data are expressed by means and standard deviation
Time Frame: Baseline and 16 Weeks
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Ankylosing Spondylitis Control | Mobility in AS | Mobility Plus Elastic Resistance Exercise in AS
Number analyzed (Participants) | 18 | 17 | 20
Centimeters
  baseline | 9.9 (2.7) | 14.2 (5.6) | 10.9 (3.6)
  16 weeks | 10.0 (2.5) | 9.5 (2.3) | 9.2 (1.6)
Statistical Analysis 1: Comparison: Ankylosing Spondylitis Control; Test type: Superiority or Other; p = 1, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mobility in AS; Test type: Superiority or Other; p = 0.000, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.350, Mixed Models Analysis
Statistical Analysis 4: Comparison: Ankylosing Spondylitis Control vs Mobility in AS; Test type: Superiority or Other; p = 0.997, Mixed Models Analysis
Statistical Analysis 5: Comparison: Ankylosing Spondylitis Control vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.970, Mixed Models Analysis
Statistical Analysis 6: Comparison: Mobility in AS vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.999, Mixed Models Analysis

13. Secondary Outcome: Tragus-coronoid Distance
Description: lateral flexion of the head (tragus-coronoid distance) was measured with a tape in centimeters. Highest score means better lateral flexion mobility of the head.Data are expressed by means and standard deviation
Time Frame: Baseline and 16 Weeks
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Ankylosing Spondylitis Control | Mobility in AS | Mobility Plus Elastic Resistance Exercise in AS
Number analyzed (Participants) | 18 | 17 | 20
Centimeters
  baseline | 9.9 (2.7) | 12.3 (4.0) | 9.7 (3.3)
  16 weeks | 10.1 (2.2) | 9.0 (2.0) | 8.8 (2.0)
Statistical Analysis 1: Comparison: Ankylosing Spondylitis Control; Test type: Superiority or Other; p = 0.997, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mobility in AS; Test type: Superiority or Other; p = 0.000, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.503, Mixed Models Analysis
Statistical Analysis 4: Comparison: Ankylosing Spondylitis Control vs Mobility in AS; Test type: Superiority or Other; p = 0.814, Mixed Models Analysis
Statistical Analysis 5: Comparison: Ankylosing Spondylitis Control vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.643, Mixed Models Analysis
Statistical Analysis 6: Comparison: Mobility in AS vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.999, Mixed Models Analysis

14. Secondary Outcome: Finger Floor Distance
Description: Distance between third finger of the hand and the floor while in lumbar flexion. It was measured with a tape in centimeters. Highest score means better torso flexion mobility. Data are expressed by means and standard deviation
Time Frame: Baseline and 16 Weeks
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Ankylosing Spondylitis Control | Mobility in AS | Mobility Plus Elastic Resistance Exercise in AS
Number analyzed (Participants) | 18 | 17 | 20
Centimeters
  baseline | 27.6 (13.3) | 27.1 (13.7) | 23.7 (12.0)
  16 weeks | 29.5 (13.6) | 24.2 (13.3) | 20.3 (11.8)
Statistical Analysis 1: Comparison: Ankylosing Spondylitis Control; Test type: Superiority or Other; p = 0.787, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mobility in AS; Test type: Superiority or Other; p = 0.408, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.157, Mixed Models Analysis
Statistical Analysis 4: Comparison: Ankylosing Spondylitis Control vs Mobility in AS; Test type: Superiority or Other; p = 0.835, Mixed Models Analysis
Statistical Analysis 5: Comparison: Ankylosing Spondylitis Control vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.256, Mixed Models Analysis
Statistical Analysis 6: Comparison: Mobility in AS vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.935, Mixed Models Analysis

15. Secondary Outcome: Chest Expansion
Description: Chest expansion was measured with a tape in centimeters between inspiration and breathing exhaling. Highest score means better chest expansion. Data are expressed by means and standard deviation.
Time Frame: Baseline and 16 Weeks
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Ankylosing Spondylitis Control | Mobility in AS | Mobility Plus Elastic Resistance Exercise in AS
Number analyzed (Participants) | 18 | 17 | 20
Centimeters
  baseline | 2.8 (1.3) | 2.8 (1.2) | 3.6 (1.7)
  16 weeks | 3.0 (1.9) | 3.3 (1.2) | 4.3 (1.9)
Statistical Analysis 1: Comparison: Ankylosing Spondylitis Control; Test type: Superiority or Other; p = 0.978, Mixed Models Analysis
Statistical Analysis 2: Comparison: Mobility in AS; Test type: Superiority or Other; p = 0.169, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis
Statistical Analysis 4: Comparison: Ankylosing Spondylitis Control vs Mobility in AS; Test type: Superiority or Other; p = 0.993, Mixed Models Analysis
Statistical Analysis 5: Comparison: Ankylosing Spondylitis Control vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.105, Mixed Models Analysis
Statistical Analysis 6: Comparison: Mobility in AS vs Mobility Plus Elastic Resistance Exercise in AS; Test type: Superiority or Other; p = 0.335, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: during 16 weeks
Description: A baseline evaluation was done and another after 16 weeks
Arm/Group | Ankylosing Spondylitis Control | Stretching in AS | Elastic Resistance Exercise in AS
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/20
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No